CLINICAL TRIAL: NCT05650190
Title: Spectacle Lenses Visual Acuity Assessments Study
Brief Title: Spectacle Lens Visual Acuity Assessments Study
Acronym: CEDAR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SightGlass Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPRO-2209-001
Record Dates: First submitted 2022-11-28; First posted 2022-12-14 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Myopia; Myopia Progression; Juvenile Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Test Arm (Experimental): Single vision, impact resistant spectacle lenses; Test Arm
  Interventions: Device: Novel spectacle lens design
- Control Arm (Placebo Comparator): Single vision, impact resistant spectacle lenses; Control Arm
  Interventions: Device: Spectacle lenses

INTERVENTIONS:
Device: Novel spectacle lens design — Use of single vision, impact resistant spectacle lenses may reduce the rate of progression of juvenile myopia
  Arms: Test Arm
Device: Spectacle lenses — Single vision, impact resistant spectacle lenses
  Arms: Control Arm

SUMMARY:
This is a two-arm parallel group, non-dispensing study. Participants will be existing active CYPRESS Extension (CPRO-1802-002) subjects. Subjects will undergo additional visual performance assessments.

ELIGIBILITY:
Inclusion Criteria:

* Existing subject from the CYPRESS Extension study (CPRO-1802-002)
* Ability to comply with study assessments
* The subject's parent(s) or legal guardian(s) must read, understand and sign the Statement of Informed Consent and receive a fully executed coy of the form

Exclusion Criteria:

* Any current ocular infection, inflammation or irritation likely to affect vision

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2022-12-08 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Visual Acuity | 15 minutes
  Reading Speed (maximum words per minute)

SECONDARY OUTCOMES:
Near Visual Acuity with Glare | 15 minutes
  Mean and Standard Deviation at 15 minutes (short duration test)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Sabal Eye Care, Longwood, Florida
  - Kannarr Eye Care, Pittsburg, Kansas
  - Advanced Eyecare PC, Raytown, Missouri
  - SUNY School of Optometry, New York, New York
  - Vision Optique, Houston, Texas
  - William J Bogus, OD, FAAO, Salt Lake City, Utah